CLINICAL TRIAL: NCT01788748
Title: Evaluation of Fractional Bipolar Radiofrequency, and Bipolar Radiofrequency Potentiated by Infrared, in Monotherapy or Combined, for the Treatment of Striae
Brief Title: Evaluation of Fractional Bipolar Radiofrequency for the Treatment of Striae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Candela France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRB-E2VER02; 2012-A01427-36 (Other: ANSM (French health committee)); 12.084 (Other: CPP Sud Méditerranée V (ethics committee))
Record Dates: First submitted 2013-02-05; First posted 2013-02-11 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Striae
Keywords: fractional; bipolar; radiofrequency; striae; infrared; combined
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- bipolar radiofrequency and infrared (Active Comparator): The abdomen of each patient will be divided in four quadrants around the navel. One quadrant, selected randomly at the subject enrollment, will receive only bipolar radiofrequency potentiated by infrared, 3 treatments one month apart.
  Interventions: Device: bipolar radiofrequency and infrared
- fractional bipolar radiofrequency (Active Comparator): The abdomen of each patient will be divided in four quadrants around the navel. One quadrant, selected randomly at the subject enrollment, will receive only fractional bipolar radiofrequency , 3 treatments one month apart.
  Interventions: Device: fractional bipolar radiofrequency
- combined treatment (Active Comparator): The abdomen of each patient will be divided in four quadrants around the navel. One quadrant, selected randomly at the subject enrollment, will receive first bipolar radiofrequency potentiated by infrared, followed in the same session by fractional bipolar radiofrequency, 3 treatments one month apart.
  Interventions: Device: bipolar radiofrequency and infrared; Device: fractional bipolar radiofrequency

INTERVENTIONS:
Device: bipolar radiofrequency and infrared
  Other Names: Applicator Sublime on the platform eTwo
  Arms: bipolar radiofrequency and infrared; combined treatment
Device: fractional bipolar radiofrequency
  Other Names: applicator Sublative, platform eTwo
  Arms: combined treatment; fractional bipolar radiofrequency

SUMMARY:
This is an interventional open prospective randomized study, done in two sites.

The main purpose of this study is to evaluate the efficacy of the combination of bipolar radiofrequency potentiated by an infrared light followed by fractional bipolar radiofrequency for the treatment of striae on the abdomen.

In order to have a more complete and accurate study, each technology will also be evaluated separately. This will allow the comparison of the effect of each treatment, in monotherapy or combined.

DETAILED DESCRIPTION:
Stria is a very common condition that affects psychologically and aesthetically a lot of patients. It is a linear atrophic scar. So, to be treated, it needs to have both a superficial and a deep impact.

Several technologies have already been tested for this indication, but none of them have been proved at the same time effective and without a high risk of side effects for all skin types. As radiofrequency is an electrical current, it is not absorbed and does not see melanin. So it can be used on all skin types.

When using fractional bipolar radiofrequency, the current goes from small electrodes to return electrodes. Around the small electrodes appear some epidermal ablation, coagulation and deeper thermal damage. This means it has a superficial and a deep effect.

Using infrared combined with bipolar radiofrequency allows the infrared to pre-heat the skin so as to help the radiofrequency to go deeper in the skin more easily. This has a deep effect in the dermis.

In this study, both technologies will be used. At least 20 patients will be treated in two different sites.

The abdomen of each patient will be divided in four quadrants around the navel. Each quadrant will receive a total of three treatments one month apart:

* One quadrant will be the control (no treatment will be done)
* One quadrant will receive each time only bipolar radiofrequency potentiated by infrared
* One quadrant will receive each time only fractional bipolar radiofrequency
* One quadrant will receive each time first bipolar radiofrequency potentiated by infrared, followed in the same session by fractional bipolar radiofrequency.

The choice of the treatment for each area will be randomized at the enrollment of the patient in the study.

There will be two follow-up sessions 3 and 6 months after the last treatment.

The evaluation will be done mainly by 3D acquisitions. This will allow measuring the length, width and depth of the striae and evaluating their evolution after the treatment.

Some patients, if they agree, will also have in vivo confocal microscopy before the first treatment and 6 months after the last one. This will give more information on the collagen and elastin changes.

Four patients, who accept it, will have biopsies performed before the first treatment and 6 months after the last one to also show the evolution of the skin structure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subject over 18 years old, with striae on all the abdomen (white or red)
* Consent form signed by subjects
* Affiliation to social security

Exclusion Criteria:

* Electrical implants (pace maker, defibrillator) or superficial metallic implants (gold thread…)
* Pregnant woman
* Woman who can procreate without using an effective birth control
* Deficient immune system due to immunosuppressive diseases such as AIDS or HIV, or use of immunosuppressive drugs,
* Stretch marks resulting from treatment with steroids,
* Treatment with oral retinoids ongoing or stopped less than a year ago, or photosensitizing ongoing or stopped less than 3 months ago
* History of diseases stimulated by heat (recurrent herpes) on the treatment area
* Procedure less than 6 months ago performed on the treatment area,
* History of keloid scarring or difficulty in healing,
* History of allergy to xylocaine (for subjects who will have biopsy)
* Dermatological disorder requiring systemic therapy or local therapy in the area under study,
* Systemic disease in evolution (cancer or history of cancer, heart disease, uncontrolled diabetes, pain syndrome, history of neuropathy)
* Problem of coagulation and / or anticoagulant therapy,
* Vascular lesions or tattoos on the treatment area,
* Vulnerable Person: minor, under protection, deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change of striae volume | before the first treatment, 3 and 6 months after the last treatment. Months 0, 5 and 8
  The stretch marks in each area will be evaluated with a 3D camera (Antera 3D, Miravex). This will give access to the length, width and depth of each stria. Those measurements will then be compared so as to evaluate each technology.

SECONDARY OUTCOMES:
Observation of the skin structure changes with in vivo confocal microscopy | 5 months
  In vivo confocal microscopy acquisitions will be done on all subjects who agree to do so. It is a non-invasive imaging procedure that shows the different structures of the skin (such as collagen fibers and elastin). This will allow us to assess the effect of both technologies, used in monotherapy or combined, on those structures.
Observation of the skin structure changes with in vivo confocal microscopy | 8 months
  In vivo confocal microscopy acquisitions will be done on all subjects who agree to do so. It is a non-invasive imaging procedure that shows the different structures of the skin (such as collagen fibers and elastin). This will allow us to assess the effect of both technologies, used in monotherapy or combined, on those structures.
Observation of the skin structure changes by histology | 8 months
  For four patients, who previously agreed to do so, 3 biopsies will be done (one on each quadrant that will receive a treatment) before any treatment and at the 6 month follow-up session. They will be analyzed in the anatomopathology laboratory of the Archet II hospital. It will show the entire dermal and epidermal evolution after each type of treatment.
Pain assessment | 1 month
  Pain will be assessed with an analogical visual scale.
Pain assessment | 2 months
  Pain will be assessed with an analogical visual scale.
Global satisfaction | 1 month
  The global satisfaction of both the subject and the investigator will be assessed with an analogical visual scale.
Global satisfaction | 2 months
  The global satisfaction of both the subject and the investigator will be assessed with an analogical visual scale.
Double blinded pictures observation | 5 months
  Standardized pictures will be taken at the beginning of each session. Two external doctors will evaluate each picture on a Physician Global Assessment scale, without knowing to which session or to which subject it corresponds.
Double blinded pictures observation | 8 months
  Standardized pictures will be taken at the beginning of each session. Two external doctors will evaluate each picture on a Physician Global Assessment scale, without knowing to which session or to which subject it corresponds.
global satisfaction | 5 months
  The global satisfaction of both the subject and the investigator will be assessed with an analogical visual scale.
Global satisfaction | 8 months
  The global satisfaction of both the subject and the investigator will be assessed with an analogical visual scale.
Pain assessment | first day
  Pain will be assessed with an analogical visual scale.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Passeron, Pr, Principal Investigator — Hopital Archet II, service de Dermatologie
Locations (2):
- France (2):
  - Aesthetics, Bordeaux
  - CHU Archet II, Service de Dermatologie, Nice